CLINICAL TRIAL: NCT00615836
Title: A Multi-Center Extension Study Investigating the Long Term Efficacy and Safety of a Fast-Dissolving ("Melt") Formulation of Desmopressin for the Treatment of Nocturia in Adults
Brief Title: An Extension Study Investigating the Efficacy and Safety of a Fast-Dissolving ("Melt") Formulation of Desmopressin for the Treatment of Nocturia in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE992026 CS31
Record Dates: First submitted 2008-01-18; First posted 2008-02-14 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-11

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Desmopressin Melt 10 μg (Experimental): Participants received desmopressin melt 10 μg once a day, placed under the tongue one hour before bedtime until they were re-randomized to one of the other doses of desmopressin Melt (25 μg, 50 μg, or 100 μg).
  Interventions: Drug: Desmopressin Melt
- Desmopressin Melt 25 μg (Experimental): Participants received desmopressin melt 25 μg once a day, placed under the tongue one hour before bedtime for up to 2 years and 2.5 months.
  Interventions: Drug: Desmopressin Melt
- Desmopressin Melt 50 μg (Experimental): Participants received desmopressin melt 50 μg once a day, placed under the tongue one hour before bedtime for up to 2 years and 2.5 months.
  Interventions: Drug: Desmopressin Melt
- Desmopressin Melt 100 μg (Experimental): Participants received desmopressin melt 100 μg once a day, placed under the tongue one hour before bedtime for up to 2 years and 2.5 months.
  Interventions: Drug: Desmopressin Melt

INTERVENTIONS:
Drug: Desmopressin Melt — An orally disintegrating tablet of desmopressin administered under the tongue (sublingually), without water.
  Other Names: Minirin® Melt; Nocturin®; FE992026

SUMMARY:
The purpose of this study was to investigate the long term efficacy and safety of several doses of the Melt formulation of desmopressin in a broad population of adult patients with nocturia.

DETAILED DESCRIPTION:
FE992026 CS31 was a multicenter open-label extension study for patients who were enrolled in Study FE992026 CS29 (NCT00477490) and had completed at least Visit 3E in Part II of that study.

The CS29 study was structured into 2 double-blind parts (Part I and Part II). In Part I, the initial 28-day treatment period, participants were randomly assigned to 1 of 5 treatment groups: placebo or desmopressin Melt 10 μg, 25 μg, 50 μg, or 100 μg. Immediately upon completion of Part I of the study, all participants on active treatment continued into Part II on the same treatment for approximately 1 to 6 months. Participants assigned to placebo in Part I were randomly assigned to 1 of the 4 active treatments in Part II, based on re-randomization predetermined at the initial randomization (to maintain the blind). Part II began at the final visit for Part I and continued until the database for Part I was locked. Therefore, treatment duration for Part II varied between 1 and 6 months, depending upon when the participant entered.

Upon completion of Part II of CS29, participants were given the option to participate in the open-label extension study (CS31). During CS31, each participant assigned to the 10 μg dose was switched to a higher dose in an open-label manner among the remaining 3 higher doses.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to the performance of any study-related activity.
* Was randomized into Part II of Protocol FE992026 CS29 (NCT00477490), entitled "A Randomized, Double Blind,Placebo Controlled, Parallel Group, Multi-Center Study with a Double Blind Extension Investigating the Efficacy and Safety of a Fast-Dissolving ("Melt") Formulation of Desmopressin for the Treatment of Nocturia in Adults" and have completed at least Visit 3E in Part II (Day 15).

Exclusion Criteria:

* Patients using loop diuretics (furosemide, torsemide, ethacrynic acid).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2007-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (73):
- United States (64):
  - Radiant Research, Scottsdale, Arizona
  - Arkansas Primary Care Clinic, PA, Little Rock, Arkansas
  - Advanced Urology Medical Center, Anaheim, California
  - Impact Clinical Trials, Beverly Hills, California
  - California Professional Research, Newport Beach, California
  - San Diego Uro-Reseach, San Diego, California
  - Radiant Research, Santa Rosa, California
  - West Coast Clinical Research, Tarzana, California
  - Western Clinical Research, Torrance, California
  - Urology Associates PC, Denver, Colorado
  - Downtown Women's Health Care, Denver, Colorado
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Connecticut Clinical Research Center, LLC, Middlebury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Women's Health Research Group, LLC, Clearwater, Florida
  - Radiant Research - St. Petersburg, Pinellas Park, Florida
  - Sunrise Medical Research, Plantation, Florida
  - Radiant Research, Stuart, Florida
  - Tampa Bay Urology, Tampa, Florida
  - Radiant Research, West Palm Beach, Florida
  - Southeastern Medical Research Institute, Columbus, Georgia
  - Investigational site, Dunwoody, Georgia
  - Radiant Research, Inc, Chicago, Illinois
  - Accelovance, Peoria, Illinois
  - Radiant Research, Kansas City, Overland Park, Kansas
  - Benchmark Research, Metairie, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - FutureCare Studies, Inc., Springfield, Massachusetts
  - Radiant Research, Minneapolis, Edina, Minnesota
  - Radiant Research, Inc., St Louis, Missouri
  - Women's Clinic of Lincoln, P.C., Lincoln, Nebraska
  - Sheldon J Freedman Ltd, Las Vegas, Nevada
  - Central Jersey Medical Research Center, Elizabeth, New Jersey
  - Lawrenceville Urology, P.A. DBA, Lawrenceville, New Jersey
  - Urology Group of New Mexico, PC, Albuquerque, New Mexico
  - Investigational site - Adult & Pediatric Urology, Carmel, New York
  - AccuMed Research Associates, Garden City, New York
  - University Urology Associates, New York, New York
  - Upstate Urology, New York, New York
  - Hudson Valley Urology, PC, Poughkeepsie, New York
  - PharmQuest, Greensboro, North Carolina
  - New Hanover Medical Research, Wilmington, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Radiant Research Inc., Cincinnati, Ohio
  - Radiant Research - Akron, Mogadore, Ohio
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Philadelphia Clinical Research, LLC, Philadelphia, Pennsylvania
  - Advanced Clinical Concepts, West Readings, Pennsylvania
  - Radiant Research, Greer, Greer, South Carolina
  - Palmetto Medical Research, Mt. Pleasant, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Advanced Research Associates, Corpus Christi, Texas
  - Investigational site - NationsMed Clinical Research, Houston, Texas
  - Accelovance, Houston, Texas
  - Regional Medical Center and Diagnostic, Humble, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Radiant Research San Antonio, San Antonio, Texas
  - IMED Research, P.A., San Antonio, Texas
  - NationsMed, Stafford, Texas
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia PC, Virginia Beach, Virginia
  - Women's Clinical Research Center, Seattle, Washington
  - Seattle Urology Research Center, Seattle, Washington
- Canada (9):
  - Southern Interior Medical Research Inc., Kelowna, British Columbia
  - Can-Med Clinical Research Inc., Victoria, British Columbia
  - Investigational site - Clinical Research, Victoria, British Columbia
  - Investigational site - Professional Corporation, Fredericton, New Brunswick
  - The Male/Female Health and Research, Barrie, Ontario
  - Brantford Urology Research, Brantford, Ontario
  - Guelph Urology Associates, Guelph, Ontario
  - Investigational site, North Bay, Ontario
  - The Fe/Male Health Centres, Oakville, Ontario

REFERENCES:
- [Derived] Juul KV, Klein BM, Sandstrom R, Erichsen L, Norgaard JP. Gender difference in antidiuretic response to desmopressin. Am J Physiol Renal Physiol. 2011 May;300(5):F1116-22. doi: 10.1152/ajprenal.00741.2010. Epub 2011 Mar 2. PMID 21367921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open only to participants who were enrolled in Study FE992026 CS29 (NCT00477490) and had completed at least Visit 3E in Part II (Day 15) of that study. 799 patients were randomized to treatment in CS29, and 601 patients formed the intent-to-treat population in CS29. This population was used to assess durability of effect in CS31.
Pre-assignment Details: Participants were initially assigned in a blinded manner to the same treatment dose received in Study CS29. After CS29 database lock, CS31 was unblinded, and based on the results of CS29, participants assigned to 10 μg were randomly assigned at their next scheduled visit to 25 μg, 50 μg, or 100 μg of desmopressin Melt.
Groups:
- Desmopressin Melt 10 μg: Participants received desmopressin Melt 10 μg once a day, placed under the tongue 1 hour before bedtime for between 2-7 months in Study CS29, continuing in Study CS31.
  During CS31, based on the results of CS29, participants were randomly assigned to 1 of the other doses of desmopressin Melt (25 μg, 50 μg, or 100 μg).
- Desmopressin Melt 25 μg: Participants received desmopressin Melt 25 μg once a day, placed under the tongue 1 hour before bedtime for between 2-7 months in Study CS29 and for up to 2 years and 2.5 months in Study CS31.
- Desmopressin Melt 50 μg: Participants received desmopressin Melt 50 μg once a day, placed under the tongue 1 hour before bedtime for between 2-7 months in Study CS29 and for up to 2 years and 2.5 months in Study CS31.
- Desmopressin Melt 100 μg: Participants received desmopressin Melt 100 μg once a day, placed under the tongue 1 hour before bedtime for between 2-7 months in Study CS29 and for up to 2 years and 2.5 months in Study CS31.
- Placebo: Participants took a placebo 'Melt' for 28 days to complete Part I of Study CS29. In Part II, placebo patients were randomized to 1 of the other 4 treatment arms to receive active desmopressin Melt, continuing into Study CS31.
Period: Part I of Core Study (FE992026 CS29)
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg | Placebo
Started | 163 | 158 | 158 | 160 | 160
Intent-to-treat Population | 155 (Received at least 1 dose of study drug and provided at least 1 primary efficacy measure.) | 152 (Received at least 1 dose of study drug and provided at least 1 primary efficacy measure.) | 148 (Received at least 1 dose of study drug and provided at least 1 primary efficacy measure.) | 146 (Received at least 1 dose of study drug and provided at least 1 primary efficacy measure.) | 156 (Received at least 1 dose of study drug and provided at least 1 primary efficacy measure.)
Completed | 144 | 148 | 138 | 135 | 145
Not Completed | 19 | 10 | 20 | 25 | 15
Period: Extension Study (FE992026 CS31)
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg | Placebo
Started | 141 | 144 | 132 | 137 | 0
Completed | 0 | 58 | 59 | 53 | 0
Not Completed | 141 | 86 | 73 | 84 | 0
Not completed — Adverse Event | 7 | 12 | 15 | 13 | 0
Not completed — Serum sodium ≤125 mmol/L | 1 | 0 | 3 | 3 | 0
Not completed — Use of exclusionary medication | 1 | 2 | 1 | 0 | 0
Not completed — Protocol Violation | 4 | 5 | 2 | 3 | 0
Not completed — Withdrawal by Subject | 37 | 42 | 38 | 43 | 0
Not completed — Lost to Follow-up | 10 | 14 | 5 | 10 | 0
Not completed — Other | 10 | 7 | 8 | 8 | 0
Not completed — Not reported | 6 | 4 | 1 | 4 | 0
Not completed — Re-randomized to a higher dose | 65 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic data provided for the Efficacy Analysis Dataset, which consisted of the intent-to-treat population from CS29 (all randomized patients who received at least 1 dose of study drug and provided at least 1 primary efficacy measure during Part I) who were on active treatment (i.e., placebo participants are not included).
Groups:
- Desmopressin Melt 10 μg: Participants received desmopressin Melt 10 μg once a day, placed under the tongue 1 hour before bedtime until they were re-randomized to 1 of the other doses of desmopressin Melt (25 μg, 50 μg, or 100 μg).
- Desmopressin Melt 25 μg: Participants received desmopressin Melt 25 μg once a day, placed under the tongue 1 hour before bedtime for up to 2 years and 2.5 months.
- Desmopressin Melt 50 μg: Participants received desmopressin Melt 50 μg once a day, placed under the tongue 1 hour before bedtime for up to 2 years and 2.5 months.
- Desmopressin Melt 100 μg: Participants received desmopressin Melt 100 μg once a day, placed under the tongue 1 hour before bedtime for up to 2 years and 2.5 months.
- Total: Total of all reporting groups
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg | Total
Number analyzed (Participants) | 155 | 152 | 148 | 146 | 601
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (14.41) | 62.4 (13.22) | 61.6 (11.80) | 62.1 (12.34) | 61.9 (12.97)
Age, Customized [Number; unit: participants]
  <65 years | 80 | 65 | 71 | 66 | 282
  >=65 years | 75 | 87 | 77 | 80 | 319
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 65 | 71 | 66 | 275
  Male | 82 | 87 | 77 | 80 | 326
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 123 | 120 | 119 | 111 | 473
  Black/African American | 21 | 28 | 24 | 27 | 100
  Asian | 2 | 2 | 3 | 6 | 13
  American Indian/Alaskan Native | 2 | 0 | 0 | 0 | 2
  Native Hawaiian/other Pacific Islander | 1 | 1 | 0 | 0 | 2
  Other | 6 | 1 | 2 | 2 | 11
Ethnic Origin [Number; unit: participants]
  Hispanic | 10 | 10 | 13 | 6 | 39
  Not Hispanic | 145 | 142 | 135 | 140 | 562

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Number of Nocturnal Voids
Description: Participants completed a voiding diary for 3 consecutive 24-hour periods prior to the study visit in which they recorded each nocturnal urination (void). The mean number of voids per night was the average number of voids from the 3-day diary. Baseline refers to Baseline of Study CS29 and the number of weeks represents the total exposure to study drug.
  Participants in the 10μg arm are included only until the time of dose escalation.
Time Frame: Baseline of Study CS29 and Weeks 8, 12, 20, 28, 52-56, 72-76, and 92-96.
Population: Efficacy Analysis dataset = CS29 ITT population (all randomized patients who received >=1 dose of study drug and provided >=1 primary efficacy measure during Part I) who were on active treatment. # analyzed represents baseline participants. N= indicates # of participants for whom data were also available at the post-baseline time point.
Measure: Mean (Standard Deviation); unit: nocturnal voids
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 155 | 152 | 148 | 146
nocturnal voids
  8 Weeks [N=103, 96, 92, 104] | -1.12 (1.166) | -1.30 (1.180) | -1.42 (1.278) | -1.47 (1.080)
  12 Weeks [N=85, 81, 77, 81] | -1.15 (1.151) | -1.40 (1.249) | -1.48 (1.155) | -1.73 (1.040)
  20 Weeks [N=62, 58, 64, 64] | -1.25 (1.167) | -1.61 (1.175) | -1.69 (1.167) | -1.86 (1.082)
  28 Weeks [N=63, 85, 62, 62] | -1.47 (1.389) | -1.36 (1.141) | -1.49 (1.276) | -1.81 (0.903)
  52-56 Weeks [N=45, 91, 81, 77] | -1.79 (1.291) | -1.40 (1.224) | -1.78 (1.342) | -2.14 (1.109)
  72-76 Weeks [N=0, 79, 72, 67] | NA (NA) — No participants remained in this treatment group. | -1.51 (1.253) | -1.86 (1.345) | -2.24 (1.287)
  92-96 Weeks [N=0, 68, 62, 62] | NA (NA) — No participants remained in this treatment group. | -1.39 (1.180) | -1.91 (1.359) | -2.09 (1.219)

2. Primary Outcome: Percentage of Participants With a Greater Than 33% Reduction in the Mean Number of Nocturnal Voids
Description: Percentage of participants with >33% reduction from Baseline in the mean number of nocturnal urinations per night, calculated from the 3-day voiding diary completed prior to each study visit.
  Participants in the 10μg arm are included only until the time of dose escalation.
Time Frame: Baseline of Study CS29 and Weeks 8, 12, 20, 28, 52-56, 72-76, and 92-96.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 155 | 152 | 148 | 146
percentage of participants
  8 Weeks [N=103, 96, 92, 104] | 57.3 | 63.5 | 67.4 | 68.3
  12 Weeks [N=85, 81, 77, 81] | 60.0 | 67.9 | 70.1 | 81.5
  20 Weeks [N=62, 58, 64, 64] | 56.5 | 79.3 | 76.6 | 82.8
  28 Weeks [N=63, 85, 62, 62] | 63.5 | 65.9 | 74.2 | 87.1
  52-56 Weeks [N=45, 91, 81, 77] | 75.6 | 73.6 | 71.6 | 88.3
  72-76 Weeks [N=0, 79, 72, 67] | NA — No participants remained in this treatment group. | 69.6 | 77.8 | 86.6
  92-96 Weeks [N=0, 68, 62, 62] | NA — No participants remained in this treatment group. | 63.2 | 77.4 | 88.7

3. Primary Outcome: Change From Baseline in Initial Period of Undisturbed Sleep
Description: Participants completed a sleep diary on 3 consecutive mornings prior to each study visit, from which the initial period of undisturbed sleep was calculated and averaged for the 3 days. The Initial Period of Undisturbed Sleep is the time elapsed from bedtime to either first void or morning arising minus the minutes it took to fall asleep. Baseline refers to Baseline of Study CS29 and the number of weeks represents the total exposure to study drug.
  Participants in the 10μg arm are included only until the time of dose escalation.
Time Frame: Baseline of Study CS29 and Weeks 8, 12, 20, 28, 52-56, 72-76, and 92-96.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 155 | 152 | 148 | 146
minutes
  8 Weeks [N=93, 82, 83, 90] | 77.64 (118.822) | 96.58 (112.750) | 104.72 (120.236) | 126.63 (114.501)
  12 Weeks [N=78, 69, 66, 72] | 97.57 (116.855) | 116.70 (110.738) | 118.71 (112.450) | 144.77 (116.376)
  20 Weeks [N=55, 51, 59, 58] | 94.51 (113.892) | 115.60 (105.136) | 133.66 (151.510) | 155.44 (119.185)
  28 Weeks [N=59, 80, 58, 61] | 113.60 (122.291) | 116.46 (114.475) | 101.04 (121.681) | 143.86 (114.170)
  52-56 Weeks [N=42, 88, 75, 71] | 120.91 (134.943) | 110.59 (113.658) | 121.34 (129.149) | 167.72 (118.301)
  72-76 Weeks [N=0, 77, 68, 60] | NA (NA) — No participants remained in this treatment group. | 125.21 (134.963) | 137.91 (136.870) | 200.67 (137.206)
  92-96 Weeks [N=0, 66, 56, 57] | NA (NA) — No participants remained in this treatment group. | 134.14 (172.834) | 163.31 (124.169) | 185.74 (118.865)

4. Secondary Outcome: Change From Baseline in Total Sleep Time
Description: Participants completed a sleep diary on 3 consecutive mornings prior to each study visit, from which the total sleep time was calculated and averaged for the 3 days. Baseline refers to Baseline of Study CS29 and the number of weeks represents the total exposure to study drug.
  Participants in the 10μg arm are included only until the time of dose escalation.
Time Frame: Baseline of Study CS29 and Weeks 8, 12, 20, 28, 52-56, 72-76, and 92-96.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 155 | 152 | 148 | 146
minutes
  8 Weeks [N=103, 96, 91, 104] | 13.93 (65.628) | 19.77 (71.609) | 33.17 (77.892) | 14.68 (76.679)
  12 Weeks [N=85, 81, 77, 81] | 20.66 (65.419) | 24.94 (65.785) | 30.34 (68.221) | 12.90 (73.777)
  20 Weeks [N=61, 58, 64, 64] | 12.64 (63.952) | 36.13 (67.708) | 34.01 (93.074) | 24.54 (75.385)
  28 Weeks [N=64, 85, 62, 62] | 11.12 (62.382) | 34.99 (65.342) | 33.99 (74.539) | 22.25 (69.033)
  52-56 Weeks [N=46, 91, 80, 77] | 21.09 (65.705) | 20.86 (71.695) | 25.68 (95.625) | 15.84 (77.880)
  72-76 Weeks [N=0, 80, 72, 66] | NA (NA) — No participants remained in this treatment group. | 26.44 (70.467) | 33.22 (78.286) | 19.34 (92.171)
  92-96 Weeks [N=0, 67, 61, 62] | NA (NA) — No participants remained in this treatment group. | 23.45 (65.624) | 37.33 (82.320) | 26.83 (95.183)

5. Secondary Outcome: Change From Baseline in International Consultation on Incontinence Modular Questionnaire - Nocturia (ICIQ-N) Nighttime Urination Bother Score
Description: The ICIQ-N is a self-administered 4-item questionnaire designed to assess the frequency and bother of daytime and nighttime urination. To assess nighttime urination bother, participants were asked to rate the degree of bother of nighttime urination by answering the question "Night time urination: How much does this bother you?" on a scale ranging from 0 (not at all) to 10 (a great deal). Higher numbers indicate greater bother.
  Participants in the 10μg arm are included only until the time of dose escalation.
Time Frame: Baseline of Study CS29, Week 16, Visit 12 (approximately 56-78 weeks total study time) and End of Study (up to a maximum of 35 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 155 | 152 | 148 | 146
units on a scale
  Week 16 [N=34, 42, 44, 35] | -3.68 (3.409) | -2.62 (3.695) | -3.77 (3.436) | -3.71 (3.295)
  Visit 12 [N=0, 84, 77, 67] | NA (NA) — No participants remained in this treatment group. | -2.83 (3.488) | -3.77 (3.211) | -4.12 (3.240)
  End of Study [N=17, 93, 84, 82] | -3.12 (2.934) | -2.96 (3.668) | -3.46 (3.504) | -3.62 (3.512)

6. Secondary Outcome: Change From Baseline in Nocturia Quality of Life (NQoL) Overall Score
Description: The NQoL is a self-administered 13-item questionnaire designed to assess the impact of nocturia on quality of life. It contains a sleep/energy domain (6 questions), a bother/concern domain (6 questions), and 1 global QoL question (which is not included in the overall score). The 12 core items are scored on a 0 to 4 scale, and the overall score is calculated by transforming the raw score into a 0-100 scale with higher numbers indicating better impact on quality of life.
  Participants in the 10μg arm are included only until the time of dose escalation.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 155 | 152 | 148 | 146
units on a scale
  Week 16 [N=34, 42, 44, 35] | 20.16 (29.515) | 22.42 (18.752) | 22.06 (21.985) | 26.13 (22.728)
  Visit 12 [N=0, 84, 77, 66] | NA (NA) — No participants remained in this treatment group. | 19.37 (19.362) | 21.51 (22.838) | 19.89 (19.684)
  End of Study [N=17, 94, 85, 80] | 12.87 (16.913) | 17.46 (20.497) | 19.13 (23.393) | 18.36 (19.684)

7. Secondary Outcome: Change From Baseline in NQoL Bother/Concern Domain Score
Description: The NQoL is a self-administered 13-item questionnaire designed to assess the impact of nocturia on quality of life. It contains a sleep/energy domain (6 questions), a bother/concern domain (6 questions), and 1 global QoL question. The 12 core items are scored on a 0 to 4 scale with higher numbers indicating a better quality of life. The bother/concern domain summary score is calculated by transforming the raw score into a 0-100 scale with higher numbers indicating a better impact on quality of life.
  Participants in the 10μg arm are included only until the time of dose escalation.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 155 | 152 | 148 | 146
units on a scale
  Week 16 [N=34, 42, 44, 35] | 22.43 (28.977) | 22.82 (20.083) | 23.30 (26.783) | 28.81 (27.010)
  Visit 12 [N=0, 83, 77, 66] | NA (NA) — No participants remained in this treatment group. | 18.27 (21.979) | 19.70 (23.702) | 17.11 (21.658)
  End of Study [N=17, 94, 84, 80] | 13.73 (23.047) | 14.23 (20.589) | 16.47 (25.871) | 16.25 (21.335)

8. Secondary Outcome: Change From Baseline in Nocturia Quality of Life (NQoL) Sleep/Energy Domain Score
Description: The NQoL is a self-administered 13-item questionnaire designed to assess the impact of nocturia on quality of life. It contains a sleep/energy domain (6 questions), a bother/concern domain (6 questions), and 1 global QoL question. The 12 core items are scored on a 0 to 4 scale with higher numbers indicating a better quality of life. The sleep/energy domain summary score is calculated by transforming the raw score into a 0-100 scale with higher numbers indicating a better impact on quality of life.
  Participants in the 10μg arm are included only until the time of dose escalation.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 155 | 152 | 148 | 146
units on a scale
  Week 16 [N=34, 42, 44, 35] | 17.89 (34.152) | 22.02 (20.645) | 20.83 (20.333) | 23.45 (21.534)
  Visit 12 [N=0, 85, 77, 66] | NA (NA) — No participants remained in this treatment group. | 20.20 (21.046) | 23.32 (25.311) | 22.66 (20.829)
  End of Study [N=17, 93, 84, 81] | 12.01 (18.510) | 20.30 (25.070) | 21.83 (23.884) | 20.58 (22.208)

9. Secondary Outcome: Change From Baseline in the Nocturia Quality of Life (NQoL) Global Quality of Life Score
Description: The NQoL is a self-administered 13-item questionnaire designed to assess the impact of nocturia on quality of life. It contains a sleep/energy domain (6 questions), a bother/concern domain (6 questions), and 1 global QoL question. The global QoL question is scored on a scale ranging from 0 (not at all) to 10 (a great deal). Higher numbers indicate better impact on quality of life.
  Participants in the 10μg arm are included only until the time of dose escalation.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 155 | 152 | 148 | 146
units on a scale
  Week 16 [N=34, 42, 44, 35] | 0.29 (0.799) | 0.36 (0.932) | 0.68 (0.708) | 0.26 (0.701)
  Visit 12 [N=0, 85, 77, 69] | NA (NA) — No participants remained in this treatment group. | 0.38 (1.112) | 0.48 (0.788) | 0.46 (0.867)
  End of Study [N=17, 93, 85, 81] | 0.18 (0.529) | 0.34 (0.801) | 0.47 (0.933) | 0.43 (0.851)

10. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) Global Score
Description: The PSQI is a self-administered 19-item questionnaire designed to assess sleep quality and disturbances. The 19 individual items are scored on an evenly weighted 0 to 3 scale and generate 7 component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these 7 components yields 1 global score ranging from 0 to 21. Higher numbers indicate greater sleep disturbance.
  Participants in the 10μg arm are included only until the time of dose escalation.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 155 | 152 | 148 | 146
units on a scale
  Week 16 [N=32, 39, 42, 34] | -2.41 (3.555) | -2.59 (3.507) | -3.52 (3.556) | -2.94 (3.084)
  Visit 12 [N=0, 80, 73, 65] | NA (NA) — No participants remained in this treatment group. | -1.59 (3.546) | -2.99 (3.747) | -2.66 (3.374)
  End of Study [N=16, 89, 78, 78] | -1.69 (2.387) | -2.12 (3.680) | -2.88 (4.212) | -1.54 (3.617)

11. Secondary Outcome: Change From Baseline in the Short Form-12, Version 2 (SF-12v2) Mental Component Summary Score
Description: The SF-12v2 was used to measure the impact of nocturia and lack of sleep on general quality of life. The SF-12 consists of 12 questions spanning 8 domains: physical functioning, role function-physical, role function-emotional, bodily pain, general health, vitality, social functioning, and mental health. These scales are combined to create 2 summary measures: the Physical Health Summary and Mental Health Summary. The Mental Health Summary score ranges from 0 to 100, where higher numbers indicate better quality of life.
  Participants in the 10μg arm are included only until the time of dose escalation.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 155 | 152 | 148 | 146
units on a scale
  Week 16 [N=34, 42, 44, 34] | 5.82 (7.784) | 3.84 (9.101) | 1.57 (8.910) | 4.14 (8.590)
  Visit 12 [N=0, 82, 73, 66] | NA (NA) — No participants remained in this treatment group. | 0.53 (8.167) | 1.39 (11.163) | 0.14 (8.858)
  End of Study [N=17, 91, 81, 80] | -0.49 (8.426) | 3.15 (9.929) | 1.77 (12.017) | 1.30 (9.954)

12. Secondary Outcome: Change From Baseline in the Short Form-12, Version 2 (SF-12v2) Physical Component Summary Score
Description: The SF-12v2 was used to measure the impact of nocturia and lack of sleep on general quality of life. The SF-12 consists of 12 questions spanning 8 domains: physical functioning, role function-physical, role function-emotional, bodily pain, general health, vitality, social functioning, and mental health. These scales are combined to create 2 summary measures: the Physical Health Summary and Mental Health Summary. The Physical Health Summary score ranges from 0 to 100, where higher numbers indicate better quality of life.
  Participants in the 10μg arm are included only until the time of dose escalation.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 155 | 152 | 148 | 146
units on a scale
  Week 16 [N=34, 42, 44, 34] | 1.23 (7.387) | 1.42 (7.444) | 2.62 (6.934) | 0.14 (8.900)
  Visit 12 [N=0, 82, 73, 66] | NA (NA) — No participants remained in this treatment group. | 1.35 (8.170) | 2.08 (8.879) | 2.28 (7.222)
  End of Study [N=17, 91, 81, 80] | 1.29 (4.077) | -0.02 (7.274) | 1.75 (8.794) | -0.67 (9.923)

13. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence that did not necessarily have a causal relationship with the study drug. An adverse drug reaction (ADR) was an AE evaluated by the Investigator as being probably or possibly causally related to treatment with the study drug.
  A serious AE (SAE) was any event that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or congenital anomaly/birth defect or was an important medical event that could have jeopardized the patient's safety or required medical or surgical intervention to prevent 1 of the outcomes listed above. The intensity of an AE was defined as severe if it resulted in the inability to work or perform usual activities.
Time Frame: From first dose of study drug in Study CS29 until the end of study CS31 (up to 35 months).
Population: Safety dataset included all patients who received at least 1 dose of study drug in either Study CS29 or CS31 and counted patients according to their study drug exposure; therefore patients could be included in more than 1 treatment arm. Of the 1023 patients, 799 were unique patients enrolled in CS29, 222 were re-randomized and 2 had dose decreased.
Measure: Number; unit: participants
Groups:
- Placebo: Participants took a placebo 'Melt' for 28 days to complete Part I of study CS29. In Part II, placebo patients were randomized to 1 of the other 4 treatment arms to receive active desmopressin Melt.
- Desmopressin Melt 10 μg: Participants received desmopressin Melt 10 μg once a day, in CS29 and CS31 until they were re-randomized to 1 of the other doses of desmopressin Melt (25 μg, 50 μg, or 100 μg).
- Desmopressin Melt 25 μg: Participants received desmopressin Melt 25 μg once a day, in CS29 or CS31. This group includes participants initially randomized to placebo and re-randomized at the end of CS29 Part I and participants initially receiving 10 μg re-randomized during CS31.
- Desmopressin Melt 50 μg: Participants received desmopressin Melt 50 μg once a day, in CS29 or CS31. This group includes participants initially randomized to placebo and re-randomized at the end of CS29 Part I and participants initially receiving 10 μg re-randomized during CS31.
- Desmopressin Melt 100 μg: Participants received desmopressin Melt 100 μg once a day, in CS29 or CS31. This group includes participants initially randomized to placebo and re-randomized at the end of CS29 Part I and participants initially receiving 10 μg re-randomized during CS31.
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Number analyzed (Participants) | 160 | 195 | 227 | 217 | 224
participants
  All adverse events | 81 | 149 | 188 | 187 | 190
  Deaths | 0 | 0 | 2 | 2 | 0
  Serious adverse events | 1 | 9 | 22 | 29 | 21
  AEs leading to discontinuation | 7 | 14 | 20 | 33 | 31
  Severe adverse events | 2 | 21 | 36 | 39 | 25
  Adverse drug reactions (ADRs) | 52 | 88 | 87 | 100 | 107

ADVERSE EVENTS:
Time Frame: From first dose of study drug in Study CS29 until the end of Study CS31 (up to 35 months).
Description: Safety dataset included all patients who received at least 1 dose of study drug in either Study CS29 or CS31 and counted patients according to their study drug exposure, therefore patients could be included in more than 1 treatment arm. Of the 1023 patients, 799 were unique patients enrolled in CS29, 222 were re-randomized and 2 had dose decreased.
Groups:
- Placebo: Participants took a placebo 'melt' for 28 days to complete Part I of study CS29. In Part II, placebo patients were randomized to one of the other four treatment arms to receive active desmopressin melt.
- Desmopressin Melt 10 μg: Participants received desmopressin melt 10 μg once a day, in CS29 and CS31 until they were re-randomized to one of the other doses of desmopressin Melt (25 μg, 50 μg, or 100 μg).
Arm/Group | Placebo | Desmopressin Melt 10 μg | Desmopressin Melt 25 μg | Desmopressin Melt 50 μg | Desmopressin Melt 100 μg
Serious Adverse Events (participants affected / at risk) | 1/160 | 9/195 | 22/227 | 29/217 | 21/224
Other Adverse Events (participants affected / at risk) | 64/160 | 113/195 | 147/227 | 154/217 | 146/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=160) | Desmopressin Melt 10 μg (N=195) | Desmopressin Melt 25 μg (N=227) | Desmopressin Melt 50 μg (N=217) | Desmopressin Melt 100 μg (N=224)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 1 | 4 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Left Ventricular Hypertrophy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sick Sinus Syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Spondylolisthesis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal Adhesions (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Scapula Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Shunt Malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Splenic Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/93 | 0/101 | 0/131 | 0/118 | 1/119 — Gender-specific to males; denominator is based on the male population
Adenosquamous Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Ureteric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Coordination Abnormal (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Radiculitis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0/93 | 0/101 | 1/131 | 0/118 | 1/119 — Gender-specific to males; denominator is based on the male population
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Haemopneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Knee Arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Aneurysm Ruptured (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Aortic Aneurysm Rupture (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Arterial Occlusive Disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Femoral Artery Occlusion (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=160) | Desmopressin Melt 10 μg (N=195) | Desmopressin Melt 25 μg (N=227) | Desmopressin Melt 50 μg (N=217) | Desmopressin Melt 100 μg (N=224)
Dry Mouth (Gastrointestinal disorders) | 44 | 70 | 62 | 64 | 61
Headache (Nervous system disorders) | 9 | 17 | 17 | 19 | 25
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 12 | 22 | 19 | 26
Hypertension (Vascular disorders) | 1 | 8 | 21 | 15 | 14
Nasopharyngitis (Infections and infestations) | 3 | 10 | 18 | 15 | 20
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 7 | 15 | 20 | 11
Urinary Tract Infection (Infections and infestations) | 1 | 10 | 19 | 15 | 15
Nausea (Gastrointestinal disorders) | 1 | 10 | 13 | 15 | 16
Diarrhoea (Gastrointestinal disorders) | 2 | 12 | 14 | 15 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3 | 5 | 15 | 15
Bronchitis (Infections and infestations) | 0 | 5 | 13 | 12 | 13
Fatigue (General disorders) | 2 | 13 | 4 | 8 | 7
Insomnia (Psychiatric disorders) | 1 | 8 | 7 | 13 | 13
Sinusitis (Infections and infestations) | 1 | 9 | 13 | 10 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 8 | 12 | 12
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 12 | 4 | 11
Dizziness (Nervous system disorders) | 1 | 9 | 10 | 11 | 11
Influenza (Infections and infestations) | 0 | 3 | 8 | 11 | 7
Oedema Peripheral (General disorders) | 0 | 6 | 2 | 11 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.